CLINICAL TRIAL: NCT02781610
Title: Standardized Treatment of Pulmonary Exacerbations II (STOP2)
Brief Title: Standardized Treatment of Pulmonary Exacerbations II
Acronym: STOP2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chris Goss (Other)
Collaborators: Cystic Fibrosis Foundation (Other); CF Therapeutics Development Network Coordinating Center (Network); Medical University of South Carolina (Other); University of Washington (Other)
Responsible Party: Sponsor-Investigator, Chris Goss, Professor of Medicine and Pediatrics, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STOP2-IP-15
Record Dates: First submitted 2016-05-12; First posted 2016-05-24 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Cystic Fibrosis
Keywords: Cystic fibrosis; Pulmonary exacerbation; Antibiotic; Treatment duration; Lung infection; Cystic Fibrosis Foundation; Cystic Fibrosis Foundation National Patient Registry
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ERR-10 (Other): ERR treatment duration - 10 Day Standard of care IV antibiotic(s) will be selected by the treating physician. Duration of treatment is the assigned intervention.
  Interventions: Drug: Standard of care IV antibiotic(s)
- ERR-14 (Other): ERR treatment duration - 14 Day Standard of care IV antibiotic(s) will be selected by the treating physician. Duration of treatment is the assigned intervention.
  Interventions: Drug: Standard of care IV antibiotic(s)
- NERR-14 (Other): NERR treatment duration - 14 Day Standard of care IV antibiotic(s) will be selected by the treating physician. Duration of treatment is the assigned intervention.
  Interventions: Drug: Standard of care IV antibiotic(s)
- NERR-21 (Other): NERR treatment duration - 21 Day Standard of care IV antibiotic(s) will be selected by the treating physician. Duration of treatment is the assigned intervention.
  Interventions: Drug: Standard of care IV antibiotic(s)

INTERVENTIONS:
Drug: Standard of care IV antibiotic(s) — IV antibiotics will be selected by the treating physician following standard of care. Duration of treatment is the assigned intervention.

SUMMARY:
Cystic fibrosis (CF), a life-shortening genetic disease, is marked by acute episodes during which symptoms of lung infection increase and lung function decreases. These pulmonary exacerbations are treated with varying antibiotics for varying time periods based on needs determined by individual patients, their families, and the health care providers. Cystic fibrosis pulmonary guidelines for the treatment of pulmonary exacerbation published by the Cystic Fibrosis Foundation (CFF) in 2009 provided recommendations for treatment and also identified key questions for which additional studies were needed.

A strong desire among clinicians to reduce treatment durations (and reduce cost, inconvenience, and potential toxicities) is in conflict with belief that patients not responding robustly to treatment might benefit from extending treatment.

This randomized, controlled, open-label study is designed to evaluate the efficacy and safety of differing durations of IV treatment, given in the hospital or at home for a pulmonary exacerbation in adult patients with CF.

DETAILED DESCRIPTION:
The study will assess the non-inferiority of 10 days versus 14 days treatment duration among patients who have an early robust improvement (ERR subjects) and the superiority of 21 days versus 14 days treatment duration among the subjects who do not meet the definition of ERR (non-ERR; NERR).

Subjects will undergo pulmonary function testing (spirometry) and complete a respiratory symptom score [Chronic Respiratory Infection Symptom Score (CRISS)] at initiation of IV treatment (Baseline/ Visit 1) and at Day 7-10 (Visit 2). At Visit 2, subjects will be allocated to groups ERR or NERR based on their initial clinical response as determined by the change in forced expiratory volume in 1 second (FEV1; percent of predicted) and CRISS from Baseline and then randomized to an IV treatment duration (nested within group).

ERR subjects [≥8% predicted improvement in FEV1 from Visit 1 to Visit 2 and CRISS reduction of ≥11 points from Visit 1 to Visit 2] will be randomized 1:1 to either 10 days or 14 days total IV antibiotic treatment duration. Remaining (NERR) subjects will be randomized 1:1 to receive either 14 or 21 days total IV antibiotic treatment duration. All subjects will be evaluated again at Visit 3, 14 days following scheduled completion of IV antibiotic treatment.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

* Male or female ≥18 years of age at Visit 1
* Documentation of a CF diagnosis
* Enrolled in the Cystic Fibrosis Foundation National Patient Registry (CFFNPR) prior to Visit 1 (US sites only)
* At the time of Visit 1, there is a plan to initiate IV antibiotics for a pulmonary exacerbation
* Performed spirometry at Visit 1 and Visit 2 and willing to perform spirometry at Visit 3
* Completed the CRISS questionnaire at Visit 1 and Visit 2 and willing to complete the Cystic Fibrosis Respiratory Symptoms Diary (CFRSD) questionnaire at Visit 3
* Willing to adhere to a specific treatment duration determined by initial response to treatment and subsequent randomization
* Willing to return for follow up Visit 3
* Written informed consent obtained from the subject or subject's legal representative

Exclusion Criteria:

Key Exclusion Criteria

* Previous randomization in this study
* Treatment with IV antibiotics in the 6 weeks prior to Visit 1
* Admission to the intensive care unit for current pulmonary exacerbation in the two weeks prior to Visit 2, unless admission was due to a desensitization protocol
* Pneumothorax in the two weeks prior to Visit 2
* Primary diagnosis for current hospitalization is unrelated to worsening lower respiratory symptoms (e.g., pulmonary clean out, distal intestinal obstruction syndrome (DIOS), sinusitis)
* Massive hemoptysis defined as > 250 cc in a 24 hour period or 100 cc/day over 4 consecutive days occurring in the two weeks prior to Visit 2
* Current pulmonary exacerbation thought to be due to allergic bronchopulmonary aspergillosis (ABPA)
* At Visit 1, receiving ongoing treatment with a duration of more than 2 weeks with prednisone equivalent to >10mg/day
* History of solid organ transplantation
* Receiving antimicrobial therapy to treat non-tuberculous mycobacterium (e.g., M. abscessus, M. avium complex) in the two weeks prior to Visit 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Actual)
Dates: Start 2016-06; Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Goss, MD, Principal Investigator — University of Washington; Patrick Flume, MD, Principal Investigator — Medical University of South Carolina
Locations (58):
- United States (57):
  - The Children's Hospital Alabama, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University Medical Center, Tucson, Arizona
  - UC San Diego Medical Center, La Jolla, California
  - Lucile S. Packard Children's Hospital, Palo Alto, California
  - University of California Davis, Health System, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Shands Hospital, Gainesville, Florida
  - Joe DiMaggio Children's Hospital (Adult), Hollywood, Florida
  - University of Miami, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - St. Luke's Regional Medical Center, Boise, Idaho
  - Saint Francis Medical Center, Peoria, Illinois
  - Indiana University Hospital, Indiana University Health, Indianapolis, Indiana
  - The University of Kansas Hospital, Kansas City, Kansas
  - John Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital (BCH), Boston, Massachusetts
  - University of Massachusetts Memorial Health Care (Worcester, MA), Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Detroit Medical Center; Harper University Hospital, Detroit, Michigan
  - Saint Louis University Hospital, St Louis, Missouri
  - St. Louis Washington University Adult - Barnes-Jewish Hospital, St Louis, Missouri
  - Billings Clinic, Billings, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Robert Wood Johnson University Hospital (New Brunswick, NJ), New Brunswick, New Jersey
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - The Long Island Jewish Medical Center, New Hyde Park, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Highland Hospital; Strong Memorial Hospital, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - North Carolina Children's Hospital, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina; Medical University of South Carolina Children's Hospital, Charleston, South Carolina
  - University of Texas Southwestern, Dallas, Texas
  - Baylor St. Lukes Medical Center, Houston, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Medical College of Virginia (Richmond, VA), Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Ruby Memorial Hospital, Morgantown, West Virginia
  - University of Wisconsin Hospital Center, Madison, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin
- Calgary Canada Adult CF Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McElvaney OJ, Heltshe SL, Odem-Davis K, West NE, Sanders DB, Fogarty B, VanDevanter DR, Flume PA, Goss CH. Adjunctive Systemic Corticosteroids for Pulmonary Exacerbations of Cystic Fibrosis. Ann Am Thorac Soc. 2024 May;21(5):716-726. doi: 10.1513/AnnalsATS.202308-673OC. PMID 38096105
- [Derived] Thornton CS, Caverly LJ, Kalikin LM, Carmody LA, McClellan S, LeBar W, Sanders DB, West NE, Goss CH, Flume PA, Heltshe SL, VanDevanter DR, LiPuma JJ. Prevalence and Clinical Impact of Respiratory Viral Infections from the STOP2 Study of Cystic Fibrosis Pulmonary Exacerbations. Ann Am Thorac Soc. 2024 Apr;21(4):595-603. doi: 10.1513/AnnalsATS.202306-576OC. PMID 37963297
- [Derived] Gold LS, Hansen RN, Patrick DL, Tabah A, Heltshe SL, Flume PA, Goss CH, West NE, Sanders DB, VanDevanter DR, Kessler L. Health care costs in a randomized trial of antimicrobial duration among cystic fibrosis patients with pulmonary exacerbations. J Cyst Fibros. 2022 Jul;21(4):594-599. doi: 10.1016/j.jcf.2022.03.001. Epub 2022 Mar 14. PMID 35300932
- [Derived] VanDevanter DR, Heltshe SL, Skalland M, West NE, Sanders DB, Goss CH, Flume PA. C-reactive protein (CRP) as a biomarker of pulmonary exacerbation presentation and treatment response. J Cyst Fibros. 2022 Jul;21(4):588-593. doi: 10.1016/j.jcf.2021.12.003. Epub 2021 Dec 18. PMID 34933824
- [Derived] Goss CH, Heltshe SL, West NE, Skalland M, Sanders DB, Jain R, Barto TL, Fogarty B, Marshall BC, VanDevanter DR, Flume PA; STOP2 Investigators. A Randomized Clinical Trial of Antimicrobial Duration for Cystic Fibrosis Pulmonary Exacerbation Treatment. Am J Respir Crit Care Med. 2021 Dec 1;204(11):1295-1305. doi: 10.1164/rccm.202102-0461OC. PMID 34469706
- [Derived] Holland P, Jahnke N. Single versus combination intravenous anti-pseudomonal antibiotic therapy for people with cystic fibrosis. Cochrane Database Syst Rev. 2021 Jun 23;6(6):CD002007. doi: 10.1002/14651858.CD002007.pub5. PMID 34159577

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ERR-10 | ERR-14 | NERR-14 | NERR-21
Started (Randomized to the ERR-10 or ERR-14 arm if allocated to ERR treatment group, or randomized to the NERR-14 or NERR-21 arm if allocated to NERR treatment group.) | 140 | 137 | 353 | 352
Completed (Completed last study visit (Day 25 for ERR-10 arm, Day 29 for ERR-14 arm or NERR-14 arm, and Day 36 for NERR-21 arm)) | 134 | 130 | 336 | 323
Not Completed | 6 | 7 | 17 | 29

BASELINE CHARACTERISTICS:
Population: Analysis for the ERR arms (ERR-10, ERR-14) was done on the per-protocol (PP) population. Analysis for the NERR arms (NERR-14, NERR-21) was done on the intent-to-treat (ITT) population. Caution: Analysis was not done on the combined total of all four treatment duration arms. Interpreting the total column is inappropriate for this study design.
Groups:
- Total: Total of all reporting groups
Arm/Group | ERR-10 | ERR-14 | NERR-14 | NERR-21 | Total
Number analyzed (Participants) | 107 | 107 | 353 | 352 | 919
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (6.34) | 27.1 (8.89) | 31.8 (10.52) | 31.5 (9.63) | 30.6 (9.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 53 | 192 | 171 | 462
  Male | 61 | 54 | 161 | 181 | 457
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 26 | 20 | 63
  Not Hispanic or Latino | 99 | 98 | 327 | 332 | 856
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 1 | 4
  Asian | 0 | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 7 | 17 | 32
  White | 98 | 100 | 335 | 322 | 855
  More than one race | 2 | 2 | 5 | 4 | 13
  Unknown or Not Reported | 2 | 2 | 2 | 6 | 12
Cystic Fibrosis (CF) Genotype [Count of Participants; unit: Participants]
  Delta F508 Homozygous | 46 | 55 | 171 | 174 | 446
  Delta F508 Heterozygous | 45 | 40 | 127 | 135 | 347
  Other/Unknown | 16 | 12 | 55 | 43 | 126
Forced Expiratory Volume in 1 second (FEV1) [Mean (Standard Deviation); unit: liters] | 1.9 (0.80) | 1.8 (0.83) | 1.8 (0.83) | 1.8 (0.76) | 1.8 (0.80)
FEV1 (% Predicted) Distribution [Count of Participants; unit: Participants]
  <50% | 60 | 61 | 192 | 194 | 507
  >=50% | 47 | 46 | 161 | 158 | 412
History of PEx in last year [Count of Participants; unit: Participants]
  0 - 1 | 43 | 45 | 145 | 144 | 377
  >=2 | 64 | 62 | 208 | 208 | 542
IV Antibiotic Treatment Location Prior to Randomization [Count of Participants; unit: Participants]
  Any Nights in Hospital | 92 | 90 | 265 | 266 | 713
  All at Home | 15 | 17 | 88 | 86 | 206
Systemic Corticosteroid Use [Count of Participants; unit: Participants] — Indication of systemic corticosteroids initiated on or after day of IV antibiotics start and before randomization.
  Participants
    Yes | 13 | 10 | 23 | 41 | 87
    No | 94 | 97 | 330 | 311 | 832

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in FEV1 % Predicted From Visit 1 to Visit 3 Between ERR-10 Day and ERR-14 Day
Description: Absolute change in FEV1 % predicted from baseline/visit 1 (start of IV antibiotic treatment) to last study visit/visit 3 (14 days after the end of IV antibiotic treatment).
Time Frame: Start of IV antibiotic treatment to 14 days after the end of IV antibiotic treatment
Population: Includes only participants within the ERR treatment group and per-protocol population, with FEV1 measurements at baseline and last study visit.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | ERR-10 | ERR-14
Number analyzed (Participants) | 107 | 107
percentage change | 13.30 (9.65) | 13.83 (9.94)
Statistical Analysis 1: Comparison: ERR-10 vs ERR-14; The ERR non-inferiority test was a priori designed to be conducted on the per-protocol (PP) population for 93% power assuming 2-sided alpha=0.05 with 155 PP participants per arm. Difference between ERR treatment duration arms is ERR-10 - ERR-14; Test type: Non-Inferiority — The non-inferiority margin is -3.5%; p = 0.0164, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-3.3 to 2.0]

2. Primary Outcome: Absolute Change in FEV1 % Predicted From Visit 1 to Visit 3 Between NERR-14 Day and NERR-21
Description: as for outcome 1
Time Frame: Start of IV antibiotic treatment to14 days after the end of IV antibiotic treatment
Population: Includes only participants within the NERR treatment group and intent-to-treat population, with FEV1 measurements at baseline and last study visit.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | NERR-14 | NERR-21
Number analyzed (Participants) | 331 | 322
percentage change | 3.60 (8.22) | 3.53 (7.13)
Statistical Analysis 1: Comparison: NERR-14 vs NERR-21; The NERR superiority test was a priori designed to be conducted on the Intent-to-Treat (ITT) population for 91% power to detect a 2.5% difference, assuming 2-sided alpha=0.05 with 285 ITT participants per arm. Difference between NERR treatment duration arms is NERR-21 - NERR-14; Test type: Superiority; p = 0.568, ANOVA; Adjusted for four dichotomous randomization strata; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.3 to 1.1]

3. Secondary Outcome: Change in CRISS From Visit 1 to Visit 3 Between ERR-10 Day and ERR-14 Day
Description: Absolute change in respiratory symptoms, as measured by the the Cystic Fibrosis Respiratory Symptoms Diary-Chronic Respiratory Infection Symptom Severity Score (CFRSD-CRISS), from baseline/visit 1 (start of IV antibiotic treatment) to last study visit/visit 3 (14 days after the end of IV antibiotic treatment). The Diary asks a participant to state the extent of their 8 respiratory symptoms: difficulty breathing, feverishness, tiredness, chills or sweats, coughing, coughing up mucus, tightness in the chest and wheezing. Each respiratory symptom is assigned a score from 0-4 based on the response, with zero corresponding to the absence of the symptom and four corresponding to symptom being present 'a great deal' or 'extremely'. A summed score (range from 0-24) is calculated for each participant and converted to a final score with a range of 0 to 100, where the lowest scores indicate improvement of symptoms.
Time Frame: Start of IV antibiotic treatment to14 days after the end of IV antibiotic treatment
Population: Includes only participants within the ERR treatment group and per-protocol (PP) population, with CRISS measurements at baseline and last study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ERR-10 | ERR-14
Number analyzed (Participants) | 106 | 107
score on a scale | -24.2 (13.21) | -25.3 (12.89)
Statistical Analysis 1: Comparison: ERR-10 vs ERR-14; Difference between ERR treatment duration arms is ERR-10 - ERR-14; Test type: Superiority; p = 0.546, t-test, 2 sided; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-2.4 to 4.6]

4. Secondary Outcome: Change in CRISS From Visit 1 to Visit 3 Between NERR-14 Day and NERR-21 Day
Description: as for outcome 3
Time Frame: Start of IV antibiotic treatment to14 days after the end of IV antibiotic treatment
Population: Includes only participants within the NERR treatment group and intent-to-treat (ITT) population, with CRISS measurements at baseline and last study visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NERR-14 | NERR-21
Number analyzed (Participants) | 335 | 322
score on a scale | -15.1 (13.74) | -16.7 (14.15)
Statistical Analysis 1: Comparison: NERR-14 vs NERR-21; Difference between NERR treatment duration arms is NERR-21 - NERR-14; Test type: Superiority; p = 0.140, t-test, 2 sided; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-3.7 to 0.5]

5. Secondary Outcome: Change in Weight From Visit 1 to Visit 3 Between ERR-10 Day and ERR-14 Day
Description: Absolute change in weight (kg) from baseline/visit 1 (start of IV antibiotic treatment) to last study visit/visit 3 (14 days after the end of IV antibiotic treatment).
Time Frame: Start of IV antibiotic treatment to14 days after the end of IV antibiotic treatment
Population: Includes only participants within the ERR treatment group and per-protocol (PP) population, with weight measurements at baseline and last study visit.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | ERR-10 | ERR-14
Number analyzed (Participants) | 107 | 106
kg | 1.7 (2.18) | 1.5 (2.21)
Statistical Analysis 1: Comparison: ERR-10 vs ERR-14; Difference between ERR treatment duration arms is ERR-10 - ERR-14; Test type: Superiority; p = 0.563, t-test, 2 sided; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.42 to 0.77]

6. Secondary Outcome: Change in Weight From Visit 1 to Visit 3 Between NERR-14 Day and NERR-21 Day
Description: as for outcome 5
Time Frame: Start of IV antibiotic treatment to14 days after the end of IV antibiotic treatment
Population: Includes only participants within the NERR treatment group and intent-to-treat (ITT) population, with weight measurements at baseline and last study visit.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | NERR-14 | NERR-21
Number analyzed (Participants) | 333 | 320
kg | 0.5 (2.16) | 0.8 (2.07)
Statistical Analysis 1: Comparison: NERR-14 vs NERR-21; Test type: Superiority — Difference between NERR treatment duration arms is NERR-21 - NERR-14; p = 0.083, t-test, 2 sided; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.04 to 0.61]

ADVERSE EVENTS:
Time Frame: For Serious Adverse Events (SAEs): Informed consent to final study visit (14 days after the end of IV antibiotic treatment). For all Other (Not Including Serious) AEs: Randomization to final study visit. Final study visit is Day 25 for ERR-10 arm, Day 29 for ERR-14 arm and NERR-14 arm, and Day 36 for NERR-21 arm.
Arm/Group | ERR-10 | ERR-14 | NERR-14 | NERR-21
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/137 | 0/353 | 0/352
Serious Adverse Events (participants affected / at risk) | 4/140 | 1/137 | 19/353 | 19/352
Other Adverse Events (participants affected / at risk) | 8/140 | 4/137 | 4/353 | 4/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERR-10 (N=140) | ERR-14 (N=137) | NERR-14 (N=353) | NERR-21 (N=352)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 (1) | 1 (1) | 9 (9) | 9 (10)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ERR-10 (N=140) | ERR-14 (N=137) | NERR-14 (N=353) | NERR-21 (N=352)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 8 (8) | 4 (4) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
Analysis was not done on the combined total of all four treatment duration arms. Interpreting the total column within demographics is inappropriate for this study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/10/NCT02781610/Prot_001.pdf
  • Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT02781610/SAP_000.pdf